CLINICAL TRIAL: NCT00692094
Title: Melatonin Entrainment of Elderly Blind Free-runners
Brief Title: Blind Elderly Melatonin Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eIRB 0194; R01AG021826 (NIH)
Record Dates: First submitted 2008-05-30; First posted 2008-06-06 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Blindness
Keywords: melatonin; circadian rhythms; sleep
MeSH Terms: conditions — Blindness | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Subjects will be given 0.5 mg at a time when melatonin should delay the timing of their body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Interventions: Biological: Melatonin
- 2 (Experimental): Subjects will be given 0.5 mg at a time when melatonin should advance the timing of their body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Interventions: Biological: Melatonin
- 3 (Experimental): Subjects will be given a larger dose (up to 10 mg) at a time when the melatonin should advance the timing of the body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Interventions: Biological: Melatonin
- 4 (Experimental): Subjects will be given a larger dose (up to 20 mg) at a time when the melatonin should advance the timing of the body clock. If the subject successfully responds to the treatment, the dose will be reduced gradually until the lowest effective dose is determined (down to 0.025 mg). If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Interventions: Biological: Melatonin

INTERVENTIONS:
Biological: Melatonin — 0.025 mg-0.5 mg, daily given at a time when it is expected to delay the timing of the body clock.
  Arms: 1
Biological: Melatonin — 0.025 mg - 0.5 mg, daily, at a time when melatonin should advance the timing of their body clock.
  Arms: 2
Biological: Melatonin — 0.025 mg - 10 mg, daily, at a time when melatonin should advance the timing of their body clock.
  Arms: 3
Biological: Melatonin — 0.025 mg - 20 mg, daily, at a time when the melatonin should advance the timing of the body clock.
  Arms: 4

SUMMARY:
The primary focus of this five-year study will be to optimize the melatonin dosing regimen for synchronizing the body clocks of elderly blind individuals to the 24-hour day.

DETAILED DESCRIPTION:
The investigators intend to study as many as 26 subjects through up to four melatonin treatment regimens, all of which involve a dose step-down in which the melatonin dose will be reduced gradually to find the lowest effective dose. The 4 treatment plans differ only in the start dose and the time of administration. Successfully treated subjects will enter a one-year intensive assessment of the safety and efficacy of melatonin treatment in which the subject will take the same dose for one year and complete biweekly assessments of efficacy and side-effects. The final phase of the study involves a placebo discontinuation, in which the subject's circadian rhythm will be returned to the baseline rhythm (this may take up to 6 months for some subjects).

ELIGIBILITY:
Inclusion Criteria:

* Adults 55-100 years old
* Blindness for at least one year, verified by an ophthalmologic exam
* Ability to comply with the requirements of the experimental protocol
* No clinically significant abnormalities (other than blindness) on a general physical examination
* Subjects must be competent to sign informed consent

Exclusion Criteria:

* Abnormal heart, liver or kidney function; a current Axis I psychiatric or substance abuse disorder according to the DSM-IV Manual
* A diagnosis of obstructive sleep apnea (apnea index > 10) or nocturnal myoclonus (> 10 associated arousals/hour)
* External demands that limit the ability to maintain a regular schedule, e.g., night shift work

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-08; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred J Lewy, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Sleep and Mood Disorders Lab, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Lewy AJ. Melatonin as a marker and phase-resetter of circadian rhythms in humans. Adv Exp Med Biol. 1999;460:425-34. doi: 10.1007/0-306-46814-x_51. No abstract available. PMID 10810544
- [Background] Sack RL, Brandes RW, Kendall AR, Lewy AJ. Entrainment of free-running circadian rhythms by melatonin in blind people. N Engl J Med. 2000 Oct 12;343(15):1070-7. doi: 10.1056/NEJM200010123431503. PMID 11027741
- [Background] Lewy AJ, Bauer VK, Hasler BP, Kendall AR, Pires ML, Sack RL. Capturing the circadian rhythms of free-running blind people with 0.5 mg melatonin. Brain Res. 2001 Nov 9;918(1-2):96-100. doi: 10.1016/s0006-8993(01)02964-x. PMID 11684046
- [Result] Lewy AJ, Emens JS, Lefler BJ, Yuhas K, Jackman AR. Melatonin entrains free-running blind people according to a physiological dose-response curve. Chronobiol Int. 2005;22(6):1093-106. doi: 10.1080/07420520500398064. PMID 16393710

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Melatonin: 0.025 Mg-0.5 mg (Delay Timing): Subjects will be given 0.5 mg at a time when melatonin should delay the timing of their body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Melatonin: 0.025 mg-0.5 mg, daily given at a time when it is expected to delay the timing of the body clock.
- Melatonin: 0.025 mg - 0.5 mg (Advance Timing): Subjects will be given 0.5 mg at a time when melatonin should advance the timing of their body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Melatonin: 0.025 mg - 0.5 mg, daily, at a time when melatonin should advance the timing of their body clock.
- Melatonin: 0.025 mg - 10 mg (Advance Timing): Subjects will be given a larger dose (up to 10 mg) at a time when the melatonin should advance the timing of the body clock. If the subject's body clock responds successfully to the dose, the dose will be reduced gradually until the lowest effective dose is found. If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Melatonin: 0.025 mg - 10 mg, daily, at a time when melatonin should advance the timing of their body clock.
- Melatonin: 0.025 mg - 20 mg (Advance Timing): Subjects will be given a larger dose (up to 20 mg) at a time when the melatonin should advance the timing of the body clock. If the subject successfully responds to the treatment, the dose will be reduced gradually until the lowest effective dose is determined (down to 0.025 mg). If the treatment does not work, the subject will be taken off treatment and later entered into a new treatment regimen.
  Melatonin: 0.025 mg - 20 mg, daily, at a time when the melatonin should advance the timing of the body clock.
Period: Overall Study
Arm/Group | Melatonin: 0.025 Mg-0.5 mg (Delay Timing) | Melatonin: 0.025 mg - 0.5 mg (Advance Timing) | Melatonin: 0.025 mg - 10 mg (Advance Timing) | Melatonin: 0.025 mg - 20 mg (Advance Timing)
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin: 0.025 Mg-0.5 mg (Delay Timing) | Melatonin: 0.025 mg - 0.5 mg (Advance Timing) | Melatonin: 0.025 mg - 10 mg (Advance Timing) | Melatonin: 0.025 mg - 20 mg (Advance Timing) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Circadian Phase Marker, as Measured by the Melatonin Levels in Serial Salivary and/or Plasma Samples.
Time Frame: biweekly throughout the entire study
Population: as for baseline characteristics
Arm/Group | Melatonin: 0.025 Mg-0.5 mg (Delay Timing) | Melatonin: 0.025 mg - 0.5 mg (Advance Timing) | Melatonin: 0.025 mg - 10 mg (Advance Timing) | Melatonin: 0.025 mg - 20 mg (Advance Timing)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Durability and Toxicity Side Effects Questionnaire
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Melatonin: 0.025 Mg-0.5 mg (Delay Timing) | Melatonin: 0.025 mg - 0.5 mg (Advance Timing) | Melatonin: 0.025 mg - 10 mg (Advance Timing) | Melatonin: 0.025 mg - 20 mg (Advance Timing)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Melatonin: 0.025 Mg-0.5 mg (Delay Timing) | Melatonin: 0.025 mg - 0.5 mg (Advance Timing) | Melatonin: 0.025 mg - 10 mg (Advance Timing) | Melatonin: 0.025 mg - 20 mg (Advance Timing)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analyses were not completed because, a unique provision in the American Recovery and Reinvestment Act (ARRA) of 2009 funding source unexpectedly prevented approval of a second year no-cost-extension in which completion of analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No